CLINICAL TRIAL: NCT03545984
Title: Evaluation of a Simulation Based Workshop to Enhance Learning of Insertion and Management of CSF Drainage Catheters in an Anesthesia Residency Program
Brief Title: Evaluation of a Simulation Based Workshop in an Anesthesia Residency Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Maged Argalious, MD, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 14-613
Record Dates: First submitted 2018-05-02; First posted 2018-06-06 (Actual); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-06

CONDITIONS: Cerebrospinal Fluid Drainage Catheter

STUDY DESIGN:
Intervention Model Description: Prospective randomized educational trial
Who Masked: Outcomes Assessor
Masking Description: The staff anesthesiologist evaluating a resident on spinal drain placement would NOT be aware of the resident's group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simulation-based training (Experimental): The simulation-based training during the first week of rotation involves step-by-step instructions on insertion of the CSF drainage catheter including aseptic technique, position of patient (lateral vs. sitting), site of insertion. The simulation training is done on a mannequin to simulate actual conditions. We plan to use a simulation model, which is basically a torso with the ability to palpate the back and spinous processes and use the epidural needle with loss of resistance technique with haptic feedback. The trainees would be able to actually perform the procedure on the manikin.
  Interventions: Other: Simulation-based learning
- problem based learning (Active Comparator): The residents allocated to the non-simulation group (problem based learning) receives standard educational teaching in the form of a problem based learning discussion during the first week of rotation.
  Interventions: Other: interactive problem based learning

INTERVENTIONS:
Other: Simulation-based learning — Simulation-based teaching involves using done on a mannequin to simulate actual conditions
  Other Names: Simulation
  Arms: simulation-based training
Other: interactive problem based learning — Standard teaching (problem based learning discussion) during cardiac/vascular rotation
  Other Names: PBL
  Arms: problem based learning

SUMMARY:
The study aim is to determine whether simulation based learning would improve senior anesthesiology residents' patient care performance during the insertion and management of cerebrospinal fluid drainage catheters when compared to interactive problem based learning (PBL) using the Anesthetist's Nontechnical Skills Global rating scale

DETAILED DESCRIPTION:
This prospective randomized trial allocates anesthesia residents into two educational groups and compares resident's performance on the the composite score (Anesthetist's Nontechnical Skills Global Rating Scale) assigned by supervising anesthesiologists after the insertion and management of cerebrospinal fluid drainage catheter during resident's vascular rotation.

The senior residents (CA-3 and CA-2) rotating through the vascular rotation at the Cleveland Clinic main campus starting December 2014 are randomly allocated to simulation based learning versus problem based learning using computer generated randomization. Randomization occurs prior to the start of the vascular rotation. The randomization is designed to allocate all residents (usually one or 2 residents) rotating through the vascular rotation each month (4 week rotation) to either simulation or problem based learning. The learning activity (whether simulation based or problem based) is scheduled to occur in the first week of the vascular rotation and the content of the educational activities (simulation based and problem based) is designed to cover the same educational material. Two of the authors of the study moderate all educational activities interchangeably (simulation and problem based). Simulation based learning required advanced scheduling of activities with our simulation center to ensure space and equipment availability and is a key factor in the decision to perform the randomization in 4 month intervals rather than month to month.

The primary outcome is the composite score (Anesthetist's Nontechnical Skills Global Rating Scale) received by participating residents during their first CSF drainage catheter insertion and management as evaluated by their supervising cardiothoracic anesthesiologists. Evaluating staff anesthesiologists is blinded to the residents' allocation group and were not involved in the study.

Baseline and outcomes data are prospectively collected on participating residents and respective patients undergoing thoracic aortic vascular procedures requiring CSF drainage catheters at the Cleveland Clinic main campus during the study period. Complications of CSF drainage catheters is also collected by looking into the EPIC of all the patients who had CSF drainage catheters handled by the residents in the study. Patients are followed up till they leave the hospital to evaluate if they developed any complications like paraplegia, infection, retained fragments. This will be a secondary descriptive outcome.

The simulation scenario consists of a patient requiring perioperative CSF drainage prior to undergoing thoracic aortic aneurysm surgery. The simulation involves step-by-step instructions on insertion of the CSF drainage catheter including aseptic technique, position of patient (lateral vs. sitting), site of insertion. The simulation training is done on a mannequin to simulate actual conditions. We plan to use a simulation model, which is basically a torso with the ability to palpate the back and spinous processes and use the epidural needle with loss of resistance technique with haptic feedback. The trainees would be able to actually perform the procedure on the manikin.

Various commercial CSF drainage kits are available. We will use the Medtronic lumbar drainage kit, which is available in the OR. Sterile technique, including chlorhexidine prep, full gown, sterile drape, sterile gloves, mask, hat. Insertion is typically at L3-L4 or L4-L5.The Tuohy needle will be inserted with the bevel facing cephalad in incremental fashion with loss of resistance technique until the epidural space is reached and then inserted further till a distinct pop is felt and the subarachnoid space entered. This will be confirmed by free flow of CSF from the Tuohy needle. The CSF catheter will then be inserted through the Tuohy needle, taking care to avoid marked seepage of CSF by minimizing the duration between trocar withdrawal and catheter introduction. The technique of using wire reinforced catheters as opposed to ordinary catheters will be demonstrated ( available on Integra CSF drainage catheters). The catheter will be threaded approximately 5 to 7 cm past the needle into the intrathecal space, the needle will be gently removed and the catheter secured with a clear occlusive dressing. Confirmation of free CSF drainage is obtained prior to dressing. The simulation would continue needing assembly and attachment of the catheter to the monitor through a transducer and learning how to drain the CSF at a particular preset value.

The residents allocated to the non simulation group (problem based learning) receives standard educational teaching in the form of a problem based learning discussion during the first week of rotation.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia residents in their CA-2 or CA-3 year in the vascular rotation who would need to monitor and take care of these systems as well as perform lumbar CSF drainage in the operating room (for thoracic aortic vascular procedures-open and endovascular) or cardiovascular ICU.

Exclusion Criteria:

* Anesthesia residents who already were enrolled in the study during their previous vascular rotation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maged Argalious, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Several residents who were randomized were unable to complete the study because they did not participate in the management of patients undergoing open or endovascular aortic surgery that required CSF drainage catheter insertion during their rotation..
Pre-assignment Details: This educational randomized trial was conducted on residents and they were enrolled and randomized in two study groups (arms) corresponding to two educational methods. Patients were not considered enrolled in this study.
Period: Overall Study
Arm/Group | Simulation-based Training | Problem Based Learning
Started | 24 | 24
Completed | 13 | 15
Not Completed | 11 | 9
Not completed — CSF cases not present during rotation | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simulation-based Training | Problem Based Learning | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — The subjects of study - anesthesia residents. This data was not collected for anesthesia residents. | NA (NA) — The subjects of study - anesthesia residents. This data was not collected for anesthesia residents. | NA (NA) — The subjects of study - anesthesia residents. This data was not collected for anesthesia residents.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — The subjects of study - anesthesia residents. This data was not collected for anesthesia residents | NA — The subjects of study - anesthesia residents. This data was not collected for anesthesia residents | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — The subjects of study - anesthesia residents. This data was not collected for anesthesia residents | NA — The subjects of study - anesthesia residents. This data was not collected for anesthesia residents | NA — Total not calculated because data are not available (NA) in one or more arms.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — The study participants - anesthesia residents. This info not collected for study participants. | NA — The study participants - anesthesia residents. This info not collected for study participants. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | NA — The study participants - anesthesia residents. This info not collected for study participants. | NA — The study participants - anesthesia residents. This info not collected for study participants. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — The study participants - anesthesia residents. This info not collected for study participants. | NA — The study participants - anesthesia residents. This info not collected for study participants. | NA — Total not calculated because data are not available (NA) in one or more arms.
Months of training as CA3 [Mean (Standard Deviation); unit: months] | 6.8 (3.0) | 6.3 (3.4) | 6.5 (3.2)
Spinal Drain Placed in the past [Count of Participants; unit: Participants] | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Composite Staff Evaluation Score (Anesthetist's Nontechnical Skills Global Rating Scale)
Description: The composite score is a continuous outcome varies between 0 and 16; 0 being the worst possible score and 16 the best possible score. Composite score received by a resident from a supervising anesthesiologist; validated scoring system based on Anesthetist's Nontechnical Skills (ANTS) Global Rating Scale. The hierarchical ANTS scoring system consists at the highest level of four basic skill categories, namely task management, team working, situation awareness, and decision making. These skill categories are further divided up into 16 skill elements and then each "element" is scored 0-1 and then all elements are summed for a total score of 0-16. The decision to report outcome in categories (Score 14-16, Score 11-13, Score 10 and below) instead of numeric contentious outcome was data driven and not represent any specified performance categories(i.e., "best performance", "good performance", "poor performance").
Time Frame: just after first CSF drainage catheter insertion and during 4-week vascular rotation; at least by the end of 4-week rotation
Measure: Count of Participants; unit: Participants
Arm/Group | Simulation-based Training | Problem Based Learning
Number analyzed (Participants) | 13 | 15
Participants
  Score 14-16 | 10 | 11
  Score 11-13 | 2 | 4
  Score 10 and below | 1 | 0

ADVERSE EVENTS:
Time Frame: Till patients' hospital discharge, an average of 3 days
Description: Adverse events collected during this study included complications occurring due to the placement of CSF drainage catheters. Adverse events might occur during or after CSF placement procedure and were recorded for residents (study subject) who performed the procedure; next, adverse events were summarized by two study groups.
Arm/Group | Simulation-based Training | Problem Based Learning
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 4/13 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simulation-based Training (N=13) | Problem Based Learning (N=15)
Bloody tinged CSF drainage in the postop period (Injury, poisoning and procedural complications) | 1 | 2
Bloody tap during CSF catheter insertion (Injury, poisoning and procedural complications) | 2 | 1
Spinal cord ischemia/new postoperative neurological deficits (Injury, poisoning and procedural complications) | 1 | 0
Postoperative CNS infection/meningitis (Injury, poisoning and procedural complications) | 0 | 0

LIMITATIONS AND CAVEATS:
Many of the residents who were randomized in the study did not participate in the care of patients requiring cerebrospinal fluid drainage catheters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03545984/Prot_SAP_000.pdf